CLINICAL TRIAL: NCT06917378
Title: The Multicenter Study to Evaluate Clinical and Angiographic Factors in Patients With Coronary Artery Chronic Total Occlusion in Taiwan
Brief Title: TRIO CTO (Taiwan Research Initiative on Coronary Total Occlusion)
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Chang Gung Memorial Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Hsien-Li Kao, Director of Cardiovascular Center, National Taiwan University Hospital
Other Study IDs: 202409095RINC
Record Dates: First submitted 2024-10-24; First posted 2025-04-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2024-10

CONDITIONS: Chronic Total Occlusion (CTO)
Keywords: CTO; Coronary Chronic Total Occlusion; Coronary artery disease; Coronary intervention; Collateral channel
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Successful CTO intervention: Successful CTO intervention, subgrouped by strategies, ex. antegrade or retrograde approach
  Interventions: Procedure: Percutaneous coronary intervention of coronary chronic total occlusion
- Failed CTO intervention: Failed CTO intervention, subgrouped by strategies, ex. antegrade or retrograde approach
  Interventions: Procedure: Percutaneous coronary intervention of coronary chronic total occlusion
- No CTO intervention: CTO was not intervened

INTERVENTIONS:
Procedure: Percutaneous coronary intervention of coronary chronic total occlusion — Coronary CTO was identified by coronary angiography, and its revascularization was attempted by either antegrade, retrograde or both approach.
  Other Names: PCI to CTO
  Groups: Failed CTO intervention; Successful CTO intervention

SUMMARY:
Coronary chronic total occlusions (CTO) present a significant challenge in the field of interventional cardiology. These complex lesions, characterized by complete blockage of a coronary artery for a prolonged duration, often require specialized techniques and strategies to achieve successful revascularization.

DETAILED DESCRIPTION:
Using this consortium, we will establish a multicenter cohort to evaluate the clinical parameters, angiographic characteristics, interventional techniques, and clinical outcomes involved in coronary CTO intervention. 3 subprojects are listed here.

Subproject 1 intends to develop a novel algorithm integrating antegrade and retrograde scoring system to optimize the CTO intervention and determine the optimal timing for primary retrograde approach. Current algorithm for CTO intervention.

Subproject 2 aims to examine the strategies and outcomes of CTO involving bifurcations. Bifurcation CTO lesions present unique challenges due to their complex anatomy. Opening of the main vessel while preserving important branches is crucial for ensuring favorable long-term clinical prognosis. This subproject will investigate different strategies and devices employed in bifurcation CTO PCI to assess their efficacy and safety outcomes.

Subproject 3 investigates the treatment strategies for right coronary artery (RCA) CTOs with concomitant left main disease, which present a unique and intricate scenario, requiring careful consideration of revascularization strategies.

ELIGIBILITY:
Inclusion criteria

1. Over 20 years old
2. Chronic total occlusion confirmed by coronary angiography, and noted for more than 3 months

Exclusion criteria Nil

Ages: 20 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Over 20 years old
  2. Chronic total occlusion confirmed by coronary angiography, and noted for more than 3 months
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with technical success of CTO revascularization | 1 day
  Successful CTO recanalization with <20% residual stenosis within the treated segment and restoration of Thrombolysis in Myocardial Infarction grade 3 antegrade flow, without side branch loss
Number of participants with collateral channel tracking success | 1 day
  retrograde guidewire crossing the CC to reach the distal cap of CTO segment.
Number of participants with major adverse cerebral cardiovascular events | 5 years
  Death, CV death, myocardial infarction, stroke, repeat revascularization

SECONDARY OUTCOMES:
Number of participants with periprocedural myocardial infarction | 1 day
  Confirmed by
Number of participants with periprocedural complications | 1 day
  Periprocedural myocardial infarction, vessel perforation, stroke, urgent or emergent revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Hsien-Li Kao, MD, Principal Investigator — National Taiwan University Hospital
Locations (3):
- Taiwan (3):
  - Chang Gung Memorial Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossello X, Pujadas S, Serra A, Bajo E, Carreras F, Barros A, Cinca J, Pons-Llado G, Vaquerizo B. Assessment of Inducible Myocardial Ischemia, Quality of Life, and Functional Status After Successful Percutaneous Revascularization in Patients With Chronic Total Coronary Occlusion. Am J Cardiol. 2016 Mar 1;117(5):720-6. doi: 10.1016/j.amjcard.2015.12.001. Epub 2015 Dec 12. PMID 26747733
- [Background] Chen S, Karmpaliotis D, Redfors B, Shlofmitz E, Ben-Yehuda O, Crowley A, Mehdipoor G, Puskas JD, Kandzari DE, Banning AP, Morice MC, Taggart DP, Sabik JF 3rd, Serruys PW, Kappetein AP, Stone GW. Does an occluded RCA affect prognosis in patients undergoing PCI or CABG for left main coronary artery disease? Analysis from the EXCEL trial. EuroIntervention. 2019 Aug 9;15(6):e531-e538. doi: 10.4244/EIJ-D-19-00263. PMID 31186220
- [Background] Fefer P, Knudtson ML, Cheema AN, Galbraith PD, Osherov AB, Yalonetsky S, Gannot S, Samuel M, Weisbrod M, Bierstone D, Sparkes JD, Wright GA, Strauss BH. Current perspectives on coronary chronic total occlusions: the Canadian Multicenter Chronic Total Occlusions Registry. J Am Coll Cardiol. 2012 Mar 13;59(11):991-7. doi: 10.1016/j.jacc.2011.12.007. PMID 22402070
- [Background] Wu EB, Brilakis ES, Mashayekhi K, Tsuchikane E, Alaswad K, Araya M, Avran A, Azzalini L, Babunashvili AM, Bayani B, Behnes M, Bhindi R, Boudou N, Boukhris M, Bozinovic NZ, Bryniarski L, Bufe A, Buller CE, Burke MN, Buttner A, Cardoso P, Carlino M, Chen JY, Christiansen EH, Colombo A, Croce K, de Los Santos FD, de Martini T, Dens J, di Mario C, Dou K, Egred M, Elbarouni B, ElGuindy AM, Escaned J, Furkalo S, Gagnor A, Galassi AR, Garbo R, Gasparini G, Ge J, Ge L, Goel PK, Goktekin O, Gonzalo N, Grancini L, Hall A, Hanna Quesada FL, Hanratty C, Harb S, Harding SA, Hatem R, Henriques JPS, Hildick-Smith D, Hill JM, Hoye A, Jaber W, Jaffer FA, Jang Y, Jussila R, Kalnins A, Kalyanasundaram A, Kandzari DE, Kao HL, Karmpaliotis D, Kassem HH, Khatri J, Knaapen P, Kornowski R, Krestyaninov O, Kumar AVG, Lamelas PM, Lee SW, Lefevre T, Leung R, Li Y, Li Y, Lim ST, Lo S, Lombardi W, Maran A, McEntegart M, Moses J, Munawar M, Navarro A, Ngo HM, Nicholson W, Oksnes A, Olivecrona GK, Padilla L, Patel M, Pershad A, Postu M, Qian J, Quadros A, Rafeh NA, Ramunddal T, Prakasa Rao VS, Reifart N, Riley RF, Rinfret S, Saghatelyan M, Sianos G, Smith E, Spaedy A, Spratt J, Stone G, Strange JW, Tammam KO, Thompson CA, Toma A, Tremmel JA, Trinidad RS, Ungi I, Vo M, Vu VH, Walsh S, Werner G, Wojcik J, Wollmuth J, Xu B, Yamane M, Ybarra LF, Yeh RW, Zhang Q. Global Chronic Total Occlusion Crossing Algorithm: JACC State-of-the-Art Review. J Am Coll Cardiol. 2021 Aug 24;78(8):840-853. doi: 10.1016/j.jacc.2021.05.055. PMID 34412818
- [Background] Galassi AR, Werner GS, Boukhris M, Azzalini L, Mashayekhi K, Carlino M, Avran A, Konstantinidis NV, Grancini L, Bryniarski L, Garbo R, Bozinovic N, Gershlick AH, Rathore S, Di Mario C, Louvard Y, Reifart N, Sianos G. Percutaneous recanalisation of chronic total occlusions: 2019 consensus document from the EuroCTO Club. EuroIntervention. 2019 Jun 20;15(2):198-208. doi: 10.4244/EIJ-D-18-00826. PMID 30636678
- [Background] Huang CC, Lee CK, Meng SW, Hung CS, Chen YH, Lin MS, Yeh CF, Kao HL. Collateral Channel Size and Tortuosity Predict Retrograde Percutaneous Coronary Intervention Success for Chronic Total Occlusion. Circ Cardiovasc Interv. 2018 Jan;11(1):e005124. doi: 10.1161/CIRCINTERVENTIONS.117.005124. PMID 29311284